CLINICAL TRIAL: NCT05641779
Title: Pigtail Catheter for Drainage of (Pneumothorax/Simple Effusion) is a Effective Procedure
Acronym: pigtail
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed gamal gaber, resident, Assiut University
Other Study IDs: pigtail drainage
Record Dates: First submitted 2022-04-17; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pigtail — pigtail catheter insertion in chest in the pleural cavity

SUMMARY:
Assessment and evaluation of Pigtail application in drainage of pneumothorax and haemothorax.

DETAILED DESCRIPTION:
Chest injuries are common following blunt and penetrating trauma. Fewer than 10 per cent of blunt injuries and 15-30 per cent of penetrating injuries require surgical management1. Most can be managed with tube thoracostomy to expand the lung (pneumothorax) or to drain blood (haemothorax)2. Although tube thoracostomy is fairly effective, it can be associated with complications such as mispositioning, malfunction, or injury by insertion through the diaphragm or liver3-5. The standard tube size.

Has usuallybeen32-40Fr.Insertion of such a large -calibre tube requires a cut-down technique, can be traumatic, and is often associated with signiﬁcant pain and discomfort. Pigtail catheters, originally used by cardiologists to drain chronic pericardial effusion6, were later modiﬁed and adapted for pleural drainage7. Because of their small size and reduced trauma during placement, patients may experience signiﬁcantly decreased pain and discomfort. Pigtail catheters are frequently used in the paediatric population8-10, as well as in adult, non-traumatic situations11-17 Pigtail catheters inserted at the bedside have similar efﬁcacy to traditional chest tube.

ELIGIBILITY:
Inclusion Criteria:

* iatrogenic pneumothorax

Exclusion Criteria:

* Age less than 18 years.
* refused to participate.
* Unconscious.
* spontaneous pneumothorax.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patient full filing my inclusion criteria participate in my study
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Effective drainage of pleural effusion and pneumothorax | baseline
  Effective drainage of pleural effusion and pneumothorax by using the imaging Rhea's method . techniques (chest x-ray and ultrasound ) By measuring the pneumothorax rim and pleural effusion in centimeters . Sum of interpleural distance Read pneumothorax size from table PA and AP .

CONTACTS AND LOCATIONS:
Overall Officials: ali a wahab, profesor, Study Director — Assiut University; mahmoud h elnaby, lecturer, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Result] Chang SH, Kang YN, Chiu HY, Chiu YH. A Systematic Review and Meta-Analysis Comparing Pigtail Catheter and Chest Tube as the Initial Treatment for Pneumothorax. Chest. 2018 May;153(5):1201-1212. doi: 10.1016/j.chest.2018.01.048. Epub 2018 Feb 13. PMID 29452099